CLINICAL TRIAL: NCT02577900
Title: Randomized, Controlled Study of Nanocrystalline Silver, Manuka Honey and Conventional Dressing in Healing Diabetic Foot Ulcer
Brief Title: Diabetic Foot Ulcer Study on Topical Interventions
Acronym: DFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Tsang Ka Kit, Nurse consultant, Queen Elizabeth Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QEH-O&T-001
Record Dates: First submitted 2015-10-11; First posted 2015-10-16 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Foot
Keywords: foot ulcer and honey and silver
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acticoat absorbent (Experimental): Apply Acticoat absorbent onto the ulcer
  Interventions: Device: Acticoat absorbent
- Honey gel sheet (Active Comparator): Apply Honey gel sheet onto the ulcer
  Interventions: Device: Honey gel sheet
- Jelonet (Other): Apply Jelonet onto the ulcer
  Interventions: Device: Jelonet

INTERVENTIONS:
Device: Acticoat absorbent — Apply Acticoat absorbent daily onto diabetic foot ulcer in 12-week study interval
  Other Names: nanocrystalline silver alginate
  Arms: Acticoat absorbent
Device: Honey gel sheet — Apply Honey gel sheet daily onto diabetic foot ulcer in 12-week study interval
  Other Names: Manuka honey alginate
  Arms: Honey gel sheet
Device: Jelonet — Apply Jelonet daily onto diabetic foot ulcer in 12-week study interval
  Other Names: paraffin tulle
  Arms: Jelonet

SUMMARY:
The purpose of this study is to determine whether nanocrystalline silver dressing, manuka honey dressing and conventional dressing are effective in the treatment of diabetic foot ulcer.

DETAILED DESCRIPTION:
Patient flow The target subjects were screened in the orthopedic department of two regional hospitals and one general outpatient clinic (GOPD). Those eligible potential subjects were recruited after they discharged from hospital according to the selection criteria. All the subjects were referred and intervened in an orthopedic nurse clinic a regional hospital. The subjects were randomized into three groups through a fixed block of 10 by online software. A sequence of assignment was generated and put into a sealed envelope by a research assistant. The investigator did not involve in randomization process and allocation sequence. The subjects were enrolled and allocated to different treatment arms according to the allocation sequence.

Data collection Outcome assessor blinding was employed in this study. A research assistant was responsible for measuring the wound size and taking clinical photo. In every clinical visit, the research assistant waited outside the clinic until the removal and proper cleansing of the wound by the first author so that she unaware of the topical treatment option. The subjects would be discontinued follow up when the wound was completely healed or till the end of 12-week study period.

Intervention All participants attended the nurse clinic for follow-up by the first author (nurse consultant) weekly in the first four week and then biweekly till 12 weeks of follow up period. They were nine clinical attendances totally. At each visit, sharp debridement for the non-viable tissue and stimulation of the vascularity on the avascular tissue were performed if needed by the first author. Then, he applied the topical dressing according to randomization sequence.

Statistical analysis All the analysis will be carried out according to the intention-to-treat principle. SPSS Statistics for Mac version 22 (SPSS Inc, Chicago, Illinois) was used for data analysis. Comparison would be made among groups by Fisher's exact test for nominal data and Kruskal-Wallis test for ordinal and scale data. The complete ulcer healing was compared among groups by Kaplan-Meier estimates. General estimating equation (GEE) was used to compare the ulcer size reduction rate, the wound fluid concentration of matrix metalloproteinase -9 (MMP9), tumor necrosis factor alpha (TNF-α) and interleukin-1 alpha (IL-1α) among groups. Statistical significance was set at p < 0.05 for all tests.

Sample size calculation

* The probability of non-healing (p1) on nanocrystalline silver (nAg) group = 0.20
* The probability (p2) of non-healing on manuka honey (MH)/conventional group = 0.50
* The alpha (α) value was 0.05 and power (1-β) was 0.8
* Ratio of sample size per group was 1:1
* Therefore, the total sample subjects for 2 groups were 77. Each group needed 39 subjects. For 3 groups, the total numbers of subjects were 117.
* From the experience, 10% of patients were loss to follow up. The actual numbers of subjects needs were 129. i.e. 43 subjects per group.

Data quality assurance In order to ensure the data quality, a research assistant was assigned to verify the source document and other trial records were accurate, complete, kept up-to-date and maintained. The student investigator trained the research assistant in the data quality assurance process. The student investigator also checked the data entry sheet with raw data every month. The responsibilities of research assistant were listed as follows.

* Check the accuracy and completeness on the case screening form and consent form.
* Verify the laboratory data in the case record form (CRF) were consistent with the corresponding laboratory result.
* Verify the inter-current illness was reported on the CRF.
* Verify all withdrawals and dropouts of enrolled subjects from this trial were reported and explained on the CRF.

If there was any missing data or data inconsistency, the research assistant was clarified the data with the internal electronic record of the hospital.

Handling of missing data The nature of this study was the multiple observations of subjects in regular censored points. Thus, the missing clinical data was handled by the last observation carried forward. For those laboratory data, statistical method of general estimating equation was used for the analysis on the repeated measures among groups. The missing data was under the missing completely at random (MCAR) assumption. Therefore, the laboratory missing data did not need to make estimation in the present study.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes mellitus and
* Age 40 or above with foot ulcer and
* Ulcer with size equals or larger than 1 cm in diameter and
* Ulcer located at or below malleolar region of foot and
* Superficial ulcer, ulcer penetrates to tendon or capsule and
* Ulcer without infection, mild and moderate infection and
* Subject with no foreseeable surgery within 12-week study period

Exclusion Criteria:

* HbA1c level ≥ 10% or
* Severe ischemia with ankle-brachial index (ABI) ≤ 0.4 or
* Ulcer deep into bone and joint or
* Osteomyelitis or
* Severe ulcer infection or
* Known allergy to manuka honey/ nanocrystalline silver or
* Known case of venous ulcer or varicose vein or
* Known case of benign or malignant tumor or
* Known to have any auto-immune disease or
* A condition requiring medication that affects the immune response or
* Participation in other experimental treatment studies or
* Pregnancy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsang Ka Kit, Master, Principal Investigator — Queen Elizabeth Hospital, Hong Kong

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acticoat Absorbent | Honey Gel Sheet | Jelonet
Started | 11 | 10 | 10
Completed | 11 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acticoat Absorbent | Honey Gel Sheet | Jelonet | Total
Number analyzed (Participants) | 11 | 10 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 6 | 19
  >=65 years | 5 | 3 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.36 (11.31) | 65.6 (11.42) | 66.1 (12.31) | 64.97 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 13
  Male | 7 | 4 | 7 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Healing of Ulcer During the Observation Period
Description: The number of participants have absence of a visible wound achieved by complete epithelialization
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Acticoat Absorbent | Honey Gel Sheet | Jelonet
Number analyzed (Participants) | 11 | 10 | 10
participants | 9 | 5 | 4

2. Secondary Outcome: Change in Ulcer Size
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of ulcer size changes
Arm/Group | Acticoat Absorbent | Honey Gel Sheet | Jelonet
Number analyzed (Participants) | 11 | 10 | 10
percentage of ulcer size changes | 97.45 (5.98) | 86.25 (15.98) | 77.51 (26.40)

3. Secondary Outcome: the Change in Concentration of Matrix Metalloproteinases-9 (MMP-9) Level Inside Wound Fluid at Week 1 and Week 4
Time Frame: Week 1, Week 4
Measure: Mean (Standard Deviation); unit: ng/ ml
Arm/Group | Acticoat Absorbent | Honey Gel Sheet | Jelonet
Number analyzed (Participants) | 11 | 10 | 10
ng/ ml
  week 1 | 3412.38 (5322.27) | 5655.76 (7163.14) | 5365.84 (13725.55)
  week 4 | 5720.59 (10480.71) | 17672.54 (11276.75) | 1987.39 (2892.48)

4. Secondary Outcome: the Change in Concentration of Tumor Necrosis Factor Alpha (TNF-α) Level Inside Wound Fluid at Week 1 and Week 4
Time Frame: Week 1, Week 4
Measure: Mean (Standard Deviation); unit: ng/ ml
Arm/Group | Acticoat Absorbent | Honey Gel Sheet | Jelonet
Number analyzed (Participants) | 11 | 10 | 10
ng/ ml
  week 1 | 9.93 (6.21) | 24.89 (26.76) | 9.92 (8.83)
  week 4 | 21.77 (18.26) | 12.44 (9.13) | 11.03 (8.51)

5. Secondary Outcome: the Change in Concentration of Interleukin-1 Alpha (IL-1α) Level Inside Wound Fluid at Week 1 and Week 4
Time Frame: Week 1, Week 4
Measure: Mean (Standard Deviation); unit: ng/ ml
Arm/Group | Acticoat Absorbent | Honey Gel Sheet | Jelonet
Number analyzed (Participants) | 11 | 10 | 10
ng/ ml
  week 1 | 1.13 (1.17) | 1.93 (1.32) | 0.62 (0.71)
  week 4 | 0.57 (0.96) | 2.08 (2.28) | 2.21 (2.70)

ADVERSE EVENTS:
Arm/Group | Acticoat Absorbent | Honey Gel Sheet | Jelonet
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes